CLINICAL TRIAL: NCT03549286
Title: Assessment of Women's Insight and Understanding of Non-invasive Prenatal Testing (NIPT) During Their First Trimester Ultrasound
Brief Title: Assessment of Women's Insight and Understanding of Down's Syndrome Screening by Non-invasive Prenatal Testing (NIPT) During Their First Ultrasound
Acronym: DEPIST21
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Other Study IDs: PZ18071
Record Dates: First submitted 2018-05-25; First posted 2018-06-07 (Actual); Last update posted 2018-06-07 (Actual); Status verified 2018-05

CONDITIONS: Pregnancy
Keywords: Pregnancy; Down's syndrome; non invasive prenatal testing
MeSH Terms: conditions — Down Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- pregnant women in the first trimester ultrasound consultation: Participation in the study will be offered to all pregnant patients, presenting for their first trimester ultrasound consultation in the obstetrics and gynecology department of the University Hospital of Reims. The study includes the consultations of all the certified doctors of the Maternity Department of the Reims University Hospital carrying out the first trimester ultrasounds. It will concern all the ranges of consultation regardless of the doctor who performs the consultation.
  Interventions: Other: Questionnaire passation

INTERVENTIONS:
Other: Questionnaire passation — Questionnaires assessing general knowledge about Down's syndrome screening, specific knowledge of NIPT for Down's syndrome and patient's satisfaction about provided information.

SUMMARY:
Down's syndrome is the leading cause for mental retardation in France. Screening for this chromosomal abnormality is systematically proposed during pregnancy.

Until April 2017, prenatal screening for Down's syndrome was based on a combined screening test which included fetal ultrasound markers and maternal serum hormone levels prescribed after the first trimester ultrasound. Depending on this screening result, women that presented a higher risk of ill fetuses could benefit from invasive procedures (amniocentesis or trophoblastic biopsy) in order to have a karyotype and make certain diagnosis. The latter procedure involved risks of complications such as miscarriages, infections and water break.

A new screening procedure is available since 2017. It relies on detecting an extra 21 chromosome in cell-free DNA by a simple maternal blood test, called noninvasive prenatal screening (NIPT). This screening test is highly efficient with a detection of 99 % of fetuses affected by Down's syndrome and therefore enables practitioners to avoid 95% of invasive samples. NIPT implies to proceed to a diagnosis test as well (amniocentesis and trophoblastic biopsy) to obtain karyotype and confirm diagnosis.

Few studies show a concerning level of Down's syndrome screening general strategy. There is a clear lack of understanding of the information provided by the health professional during the first trimester ultrasound. Women report feeling uninformed and confused about French screening strategy. Nevertheless, high quality insight is essential to ensure validity of women's consent to perform Down's syndrome screening and quality of provided health care.

Since introduction of NIPT, no study has been carried out to assess women's prior knowledge to NIPT for Down's syndrome. Main objective of the study is therefore to evaluate women's information and understanding of Down's syndrome screening using NIPT. Secondary objectives stand in collecting modalities of the provided information by the doctor performing the first ultrasound and assess patient's satisfaction regarding this information.

Understanding of this new screening strategy by pregnant women is a key issue in decision making. This observational study is intended for all pregnant patients from 11 to 17 + 6 WA (weeks of amenorrhea) expecting a single baby, consulting in the obstetrics and gynecology department of the University Hospital of Reims for their 1st trimester ultrasound. Participation to the study will not change patient's medical care. The doctor who carries out the ultrasound will not be aware of the patient's participation in the study. Concordant results with literature using the experience of what was done for Down's syndrome screening prior to NIPT are expected. Communication on this matter to the lay public is scarce. Level of knowledge regarding NIPT before the consultation is expected to be insufficient. The absolute necessity of upstream information (brochure provided by secretaries, information disclosed throughout the three month pregnancy consultation, booklet delivered with initial documents ....) to enhance patient's comprehension and satisfaction will be highlighted.

DETAILED DESCRIPTION:
- Introduction

o NIPT (non invasive prenatal testing)

Down's syndrome is the leading cause of mental retardation in France. It results form in a supernumerary chromosome 21. It concerns on average of 27.3 per 10,000 pregnancies and 6.6 per 10,000 births, frequency of non-disjunctive chromosomes increasing exponentially with age. French national policy is to systematically propose Down's syndrome screening during pregnancy which is intended for supposed healthy fetuses. Purpose is to target high-risk fetuses for which a diagnosis will be proposed and make minimum number of fetal samples, to decrease on one hand risk of miscarriages for healthy fetuses as well as health care cost on the other hand.

Prenatal screening for Down's syndrome was initially based on a risk calculation from maternal serum markers (HCG and PAPP-A) combined to nuchal translucency during first trimester ultrasound and personal data (maternal age, antecedent of Down's syndrome). Diagnosis by invasive sampling was therefore only proposed to high-risk fetuses group or for fetuses with ultrasound abnormalities. This combined strategy is accounted for a sensitivity of 81.2% and a false positive rate of 2.8% with a detection probability between 73% to 100%. Invasive samples are carried out in 5% of cases and are associated with a risk of induced miscarriage of 0.5% to 1%.

Since 2017, a new screening strategy is available from extracting fetal fraction in cell-free DNA in maternal plasma from a simple blood sample. NIPT (noninvasive prenatal testing) was born form new sequencing techniques and estimates the amount of fetal free circulating DNA in maternal blood in order to detect presence of a supernumerary 21 chromosome. This technique has sensitivity and a specificity that are far superior to "classical screening" and avoids 95% of invasive sampling. A negative result makes it possible to exclude with almost complete certainty the diagnosis of Down's syndrome but must always be confirmed by a karyotype in case of a positive test. Its effectiveness in the detection of a fetal Down's syndrome is higher than classical screening. In order to reduce invasive sampling number and improve performance of screening, NIPT was included in French screening strategy in April 2017. NIPT is now proposed to pregnant women in the following indications: for pregnant women with an increased risk of Down's syndrome: combined risk result between 1/51 and 1/1 000, maternal age above 38 years old who could not benefit from serum markers and parents presenting a Robertsonian translocation involving a Down's syndrome, chromosome 21 or a history of fetal aneuploidy. NIPT is not indicated in case of ultrasound anomalies. As a screening test, it must absolutely be completed by a karyotype in case of positive and does not substitute for a diagnostic test.

o Women's insight about Down's syndrome screening

In parallel with Down's syndrome screening reform implementation in 2009, women's acknowledgement and feelings about the screening strategy were collected and revealed low awareness and lack of understanding of the risk calculations used in Down's syndrome screening. In a French study, about 21% of patients seem to confuse notion of risk calculation and diagnosis, and 64% of them do not feel well informed about the screening. This highlights flaws in the provided information on Down's syndrome screening by health care professionals. What's more, patient's knowledge of limitations of ultrasound in the diagnosis of T21 seem insufficient, putting to light confusion between screening test and diagnosis test.

Highlighting the lack of patient's screening understanding brings up the issue of validity of consent and the possibility of informed choice regarding screening. It is therefore essential for practitioners to deliver high quality information during consultations and taking the time necessary to explain screening strategy to women. Since introduction of NIPT for Down's syndrome, no studies have been conducted regarding patient information and understanding of the updated screening strategy which is provided mainly during and after the first trimester ultrasound. A recent German study conducted in high-risk population of T21 (> 1/200) shows that the majority of women have sufficient knowledge to make an informed choice.

It therefore seems important to ensure that the quality of the information delivered is sufficient during the first trimester ultrasound. French national authority (HAS) insist on guaranteeing fair access to appropriate and quality information for all pregnant women. Consequently, mentioning implication of a positive screening test results decreases anxiety, which automatically have an impact on the duration of the consultation. There is currently no French study on patient understanding and knowledge of Down's syndrome screening and NIPT testing since its formal entry as a tool in Down's syndrome screening.

- Objective

The aim of this study is to assess the quality of information and understanding of Down's syndrome by NIPT before and after the first trimester ultrasound consultation. Secondary objectives stand in collecting modalities of the provided information (time spent, substrate used), satisfaction of women on the provided information received and identifying risk factors associated with a better understanding of the screening strategy.

Understanding of this new screening strategy by pregnant women is a key issue in decision making. We seek to highlight the absolute necessity of upstream information (brochure provided by secretaries, information disclosed throughout the three month pregnancy consultation, booklet delivered with initial documents ....) to enhance patient's comprehension and satisfaction.

- Investigation plan

This is a observational study intended for all pregnant patients from 11 to 17 + 6 WA (weeks of amenorrhea) expecting a single baby, consulting in the obstetrics and gynecology department of the University Hospital of Reims for their 1st trimester ultrasound. The study includes consultations of all certified doctors of the Maternity Department of the Reims University Hospital. It will concern all ranges of consultation regardless of the doctor who performs the consultation.

Information about the study will be given to the patient when she arrives to present herself to the secretaries. Study and its implication will be explained by a doctor a dedicated room to respect the confidentiality of the collected information. When the patient agrees to participate to the protocol (no objection form), the "pre-consult survey" will be attributed. After the consultation, the post- consult survey" will be fulfilled.

The questionnaire collects: (i) demographic characteristics, (ii) awareness of NIPT, (iii) general knowledge about Down's syndrome screening, (iiii) specific knowledge of NIPT for Down's syndrome and (iiiii) patient's satisfaction about provided information. Estimation of participation will be 30 minutes in total. Participation to the study does not change the patient's care and ultrasound realization will not be affected by the patient's participation in the study. Gynecologist performing the ultrasound will not be aware of the patients participation to the protocol. The duration of the inclusion phase will be 6 months. The time required to complete these questionnaires was estimated at half an hour (additional time to the duration of the consultation for the T1 ultrasound).

Without data from the literature regarding patient information about Down's syndrome screening since the 2017 HAS guidelines and the facilitation of access to NIPD, it was pragmatically decided to include all eligible patients. Given the activity of the obstetrics and gynecology department of Reims University Hospital and the 6-month inclusion period, an inclusion of 200 patients is planned.

ELIGIBILITY:
Inclusion Criteria:

* Major
* pregnancy between 11 and 17 +6 SA
* who consults in the gynecology department of the University Hospital of Reims for the realization of the first trimester ultrasound
* have accepted to participate in the study

Exclusion Criteria:

* Minor
* presenting a twin pregnancy (because in this indication, the serum markers are not validated nor the NIPT)
* not French speaker
* having a personal or family history of Down's syndrome
* Patients for whom the measurement of craniocaudal length during the first trimester ultrasound estimates the pregnancy before 11SA or after 17 + 6 SA
* Patients for whom ectopic pregnancy is discovered during first trimester ultrasound

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All pregnant patients, presenting for their first trimester ultrasound consultation in the obstetrics and gynecology department of the University Hospital of Reims.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-05-02 (Actual); Primary Completion 2018-11-02 (Estimated); Study Completion 2019-02-02 (Estimated)

PRIMARY OUTCOMES:
knowledge about Down's syndrome screening | Day 0
  sum of the correct responses in the 10 items questionnaire assessing knowledge about Down's syndrome screening

CONTACTS AND LOCATIONS:
Locations (1):
- Damien JOLLY, Reims, France